CLINICAL TRIAL: NCT06474572
Title: Applied Forces During Neonatal Intubation With Direct and Video Laryngoscopy at Different Heights of the Resuscitation Table: a Randomized Crossover Manikin Study
Brief Title: Applied Forces During Neonatal Intubation at Different Heights of the Resuscitation Table
Acronym: IntTab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEOUNIPD5(2024)
Record Dates: First submitted 2024-05-28; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Neonatal Disease; Intubation
Keywords: Neonate; Intubation; Direct laryngoscopy; Video laryngoscopy; Forces; Simulation
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct laryngoscope and table at xiphoid level (Active Comparator): Participants will be required to intubate the manikin with a direct laryngoscope and table at xiphoid level
  Interventions: Device: Direct laryngoscope and table at xiphoid level
- Videolaryngoscope and table at xiphoid level (Active Comparator): Participants will be required to intubate the manikin with a video laryngoscope and table at xiphoid level
  Interventions: Device: Videolaryngoscope and table at xiphoid level
- Direct laryngoscope and table at umbilical level (Active Comparator): Participants will be required to intubate the manikin with a direct laryngoscope and table at umbilical level
  Interventions: Device: Direct laryngoscope and table at umbilical level
- Videolaryngoscope and table at umbilical level (Experimental): Participants will be required to intubate the manikin with a video laryngoscope and table at umbilical level
  Interventions: Device: Videolaryngoscope and table at umbilical level

INTERVENTIONS:
Device: Direct laryngoscope and table at xiphoid level — Participants will be required to intubate the manikin with a direct laryngoscope and table at xiphoid level
  Arms: Direct laryngoscope and table at xiphoid level
Device: Videolaryngoscope and table at xiphoid level — Participants will be required to intubate the manikin with a video laryngoscope and table at xiphoid level
  Arms: Videolaryngoscope and table at xiphoid level
Device: Direct laryngoscope and table at umbilical level — Participants will be required to intubate the manikin with a direct laryngoscope and table at umbilical level
  Arms: Direct laryngoscope and table at umbilical level
Device: Videolaryngoscope and table at umbilical level — Participants will be required to intubate the manikin with a videolaryngoscope and table at umbilical level
  Arms: Videolaryngoscope and table at umbilical level

SUMMARY:
The study aims to compare the applied forces during intubation of a newborn manikin with direct and video laryngoscope at different heights of the resuscitation table. Furthermore, the success at the first attempt, the intubation time and participants' opinion on the procedures were investigated.

This is an unblinded, randomized, controlled, crossover trial on the applied forces during intubation of a newborn manikin with direct and video laryngoscope at different heights of the resuscitation table.

DETAILED DESCRIPTION:
Background: Endotracheal intubation is an important life-saving procedure for critically ill neonates. Some procedure-related aspects may affect the quality of the intubation. Optimizing the relative height between patient and operator may improve intubation procedures.

Objectives: To compare the applied forces during intubation of a newborn manikin with direct and video laryngoscope at different heights of the resuscitation table. Furthermore, the success at the first attempt, the intubation time, and participants' opinions on the procedures were investigated.

Methods: This is an unblinded, randomized, controlled, crossover trial on the applied forces during intubation of a newborn manikin with direct and video laryngoscope at different heights of the resuscitation table. Participants will be Level III NICU/PICU consultants, and pediatric residents. Randomization will be performed using a computer-generated random assignment list. The primary outcome measure will be the forces applied on the neonatal manikin during the intubation. The secondary outcome measures will be the success of the first attempt, the total time of intubation, and participants' opinions about the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Level III NICU and PICU consultants, and pediatric residents

Exclusion Criteria:

* Refusal to participate

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Magnitide of applied forces (Newton) | 3 minutes
  Magnitude of forces (measured in Newton) applied to the epiglottis and the palate of the neonatal manikin during the intubation

SECONDARY OUTCOMES:
Percentage of participants achieving the intubation success at the first attempt | 30 seconds
  The success of the first attempt will be defined as the achievement of the correct positioning of the endotracheal tube in the trachea as assessed by the external observer
Total time of intubation | 3 minutes
  Time of device positioning will be calculated as the sum of the time of device positioning in all attempts, as the procedure will be repeated in case of incorrect positioning
Participant's opinions about the procedure | 12 hours
  Participants will report: their preference about table height and device; perceived difficulty using a Likert scale (1= not difficult, 5=very difficult)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans P, Shults J, Weinberg DD, Napolitano N, Ades A, Johnston L, Levit O, Brei B, Krick J, Sawyer T, Glass K, Wile M, Hollenberg J, Rumpel J, Moussa A, Verreault A, Abou Mehrem A, Howlett A, McKanna J, Nishisaki A, Foglia EE. Intubation Competence During Neonatal Fellowship Training. Pediatrics. 2021 Jul;148(1):e2020036145. doi: 10.1542/peds.2020-036145. Epub 2021 Jun 25. PMID 34172556
- [Background] Pouppirt NR, Nassar R, Napolitano N, Nawab U, Nishisaki A, Nadkarni V, Ades A, Foglia EE. Association Between Video Laryngoscopy and Adverse Tracheal Intubation-Associated Events in the Neonatal Intensive Care Unit. J Pediatr. 2018 Oct;201:281-284.e1. doi: 10.1016/j.jpeds.2018.05.046. Epub 2018 Jul 3. PMID 29980290
- [Background] Geraghty LE, Dunne EA, Ni Chathasaigh CM, Vellinga A, Adams NC, O'Currain EM, McCarthy LK, O'Donnell CPF. Video versus Direct Laryngoscopy for Urgent Intubation of Newborn Infants. N Engl J Med. 2024 May 30;390(20):1885-1894. doi: 10.1056/NEJMoa2402785. Epub 2024 May 5. PMID 38709215
- [Background] Xue FS, Li RP, Liu GP. Dynamic optimization of height relation between anaesthetist's chest and patient's face during tracheal intubation. Br J Anaesth. 2015 Feb;114(2):348-9. doi: 10.1093/bja/aeu479. No abstract available. PMID 25596228
- [Background] Gordon JK, Bertram VE, Cavallin F, Parotto M, Cooper RM. Direct versus indirect laryngoscopy using a Macintosh video laryngoscope: a mannequin study comparing applied forces. Can J Anaesth. 2020 May;67(5):515-520. doi: 10.1007/s12630-020-01583-x. Epub 2020 Mar 9. PMID 32152886
- [Derived] Cavallin F, Pasquali G, Maglio S, Villani PE, Menciassi A, Tognarelli S, Trevisanuto D. Applied forces during neonatal intubation with direct and video laryngoscopy at different bed elevations: a randomized crossover manikin study. Eur J Pediatr. 2025 Nov 5;184(12):732. doi: 10.1007/s00431-025-06524-8. PMID 41191125